CLINICAL TRIAL: NCT00239733
Title: The Safety and Efficacy of Intravenous Anti-D for the Treatment of Thrombocytopenia in Patients With HCV Infection Prior to or During Treatment With Pegylated-interferon and Ribavirin
Brief Title: Anti-D for Treating Thrombocytopenia in Adults Infected With Hepatitis C Virus With or Without HIV Co-Infection
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: failure to enroll additional subjects
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Kristen Marks, Assistant Professor, National Institute of Allergy and Infectious Diseases (NIAID)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23AI065319-01 (NIH)
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Thrombocytopenia; Hepatitis C; HIV Infections
Keywords: HIV; HCV; Hepatitis C; Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia; Hepatitis C; HIV Infections | interventions — RHO(D) antibody; gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Participants will be given anti-D in an outpatient setting. Participants will be observed for any adverse effects for 1 hour postinfusion. Some participants may require additional doses of anti-D later in the study, depending on individual response to the drug; participants may receive 1 to 6 doses of anti-D.
  Interventions: Drug: Anti-D

INTERVENTIONS:
Drug: Anti-D — 30-minute infusion administered in an outpatient setting
  Other Names: WinRho

SUMMARY:
Thrombocytopenia occurs when a person's blood has a decreased number of platelets, which are cells involved in blood clotting. This condition may lead to uncontrolled bleeding and can be fatal. Thrombocytopenia commonly occurs with hepatitis C virus (HCV) infection or as a result of standard HCV treatment. Anti-D is an antibody approved by the Food and Drug Administration (FDA) for the treatment of HIV-related thrombocytopenia. The purpose of this study is to determine the safety and effectiveness of intravenous anti-D for the treatment of thrombocytopenia in patients with HCV infection who are starting or already undergoing treatment with peginterferon alfa-2 and ribavirin. This study will recruit HCV patients both with and without HIV co-infection.

DETAILED DESCRIPTION:
Peginterferon alfa-2 with ribavirin is the current standard of care for the treatment of HCV infection; however, severe hematologic effects, including anemia, leukopenia, and thrombocytopenia, may make this treatment less than ideal for patients with HCV. Medications to prevent or treat serious neutropenia and anemia have been established and are commonly used. However, thrombocytopenia remains a barrier to the effective treatment of HCV infection in some patients. Developing a more effective treatment for thrombocytopenia for these patients would decrease the risk of serious bleeding events. It may also improve HCV treatment outcomes by preventing dose modifications or discontinuations of peginterferon alfa-2 and ribavirin due to thrombocytopenia.

Anti-D is an antibody to the Rh (D) antigen on red blood cells. When anti-D attaches to the Rh (D) antigen, immune-mediated destruction of platelets is prevented, helping to alleviate low platelet levels in people with thrombocytopenia. This study will investigate the safety and efficacy of anti-D for the treatment of thrombocytopenia in HCV patients currently on or starting standard HCV treatment. Both HIV infected and uninfected participants will be recruited for this study.

This study will last 12 weeks. Participants in this study must be either currently on peginterferon alfa-2 and ribavirin treatment or initiating such treatment at the start of the study; these two medications will not be provided by the study. At study entry, participants will be given anti-D over a 30-minute infusion in an outpatient setting. Participants will be observed for any adverse effects for 1 hour postinfusion. Some participants may require additional doses of anti-D later in the study, depending on individual response to the drug; participants may receive 1 to 6 doses of anti-D. Efficacy of anti-D treatment will be assessed by absolute change in platelet count and the ability to sustain plaletet counts greater than 50,000 cells/microL during the study. Cytokine levels will also be monitored to gain insight on how anti-D may work with cytokines in platelet survival and clearance.

Generally, study visits will occur at study entry and Weeks 1, 2, 4, 8, and 12. In patients who require additional infusions of anti-D, there will be additional visits scheduled for each additional infusion and a postinfusion visit occurring 1 week after each infusion. All study visits will include medication history and blood collection. A clinical assessment and a targeted physical exam will occur at study entry, Weeks 1 and 12, and at additional infusion and postinfusion visits, if applicable.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* HCV-infected
* Currently on treatment for HCV OR plan to begin treatment for HCV at the start of this study
* Platelet count less than 50,000 cells/microl
* Hemoglobin greater than 10 g/dl OR greater than 11 g/dl if peginterferon treatment-naive
* Red blood cells are Rh (D) antigen-positive
* Negative Coombs direct antibody test

Inclusion Criteria for HIV Infected Group:

* HIV-infected

Inclusion Criteria for HIV Uninfected Group:

* HIV-uninfected

Exclusion Criteria:

* Prior treatment with intravenous immunoglobulin (IVIG), anti-D, or other medication for the treatment of thrombocytopenia within 30 days of study entry
* Prior serious reaction to plasma products
* Absence of spleen
* Evidence of thrombotic thrombocytopenic purpura (TTP) OR cause of thrombocytopenia other than HCV infection, HCV treatment, or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M. Marks, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital (Cornell), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ware RE, Zimmerman SA. Anti-D: mechanisms of action. Semin Hematol. 1998 Jan;35(1 Suppl 1):14-22. PMID 9523745

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti-D: Participants will be given anti-D in an outpatient setting. Participants will be observed for any adverse effects for 1 hour postinfusion. Some participants may require additional doses of anti-D later in the study, depending on individual response to the drug; participants may receive 1 to 6 doses of anti-D.
  Anti-D: 30-minute infusion administered in an outpatient setting
Period: Overall Study
Arm/Group | Anti-D
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Anti-D
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 51 [32 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6
Other baseline characteristics [Count of Participants; unit: Participants]
  HIV coinfected | 1
  Cirrhosis | 5
  Decompensated Cirrhosis | 3

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Severity of Adverse Events
Time Frame: Throughout study, for up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-D
Number analyzed (Participants) | 6
Participants
  Any SAE | 3
  Post infusion reactions | 2
  Hepatic decompensation | 1
  Any Hyperbilirubinemia | 6
  Gr 3-4 Hyperbilrubinemia | 1
  Anemia (all grade 1) | 5
  Fatigue | 4
  Fever | 2
  Dyspnea on exertion | 3
  Headache (all grade 1) | 2
  Depression (mild) | 1
  hypothyroidism | 1
  Neutropenia (likely sec to IFN) | 4
  Hospitalized | 3
  Death | 1

2. Primary Outcome: Absolute Change in Platelet Count From Baseline
Time Frame: Through Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-D
Number analyzed (Participants) | 6
Participants
  Platelet response >50,000/ul week 1 | 1
  Platelet response >50,000/ul week 2 | 2
  Platelet response >50,000/ul week 4 | 2
  Platelet response >50,000/ul week 8 | 3
  Platelet response >50,000/lu week 12 | 0
  Tp-related dose interruption peginterferon/ribavir | 1
  Anemia-related dose interruption peginterferon | 2
  Anemia-related dose interruption ribavirin | 5

ADVERSE EVENTS:
Arm/Group | Anti-D
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-D (N=6)
Hepatic decompensation (Hepatobiliary disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Seixzure/meningitis (Nervous system disorders) | 1 (1)
Death (sepsis_ (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-D (N=6)
Post infusion reactions (Vascular disorders) | 2 (2)
Hyperbilirubinemia Gr 3-4 (Hepatobiliary disorders) | 1 (1)
Anemia Gr 1 (Blood and lymphatic system disorders) | 5 (5)
Dyspnea on exertion (Cardiac disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No